CLINICAL TRIAL: NCT05986136
Title: Activation of Autophagy and Suppression of Apoptosis by Dapagliflozin Attenuates Inflammatory Bowel Disease
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tanta 1234
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Mesalamine; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Control group ( Mesalamine group, n =30 ) who will receive 1 g mesalamine three times daily for 6 months
  Interventions: Drug: Mesalamine
- Dapagliflozin group (Active Comparator): Patients will receive 1 g mesalamine three times daily plus dapagliflozin 10 mg once daily for 6 months
  Interventions: Drug: Mesalamine; Drug: Dapagliflozin 10mg Tab

INTERVENTIONS:
Drug: Mesalamine — Mesalamine, also known as 5-aminosalicylic acid (5-ASA), is a medication used to treat ulcerative colitis. It is usually used to induce or maintain remission of mildly to moderately active ulcerative colitis
Drug: Dapagliflozin 10mg Tab — Dapagliflozin has emerged as a selective SGLT2 inhibitor for the management of type-2 diabetes mellitus with minimal risk of hypoglycemia and it exerts diuretic-like actions and lowering of blood pressure, thereby, reducing the risk of hospitalization in type-2 diabetic patients with co-existing heart failure
  Arms: Dapagliflozin group

SUMMARY:
The inflammatory bowel diseases (IBD) are described as complex, recurrent inflammatory conditions which are manifested as Crohn's disease (CD) and ulcerative colitis (UC). The common symptoms of IBD include debilitating/severe diarrhea, abdominal pain, weight loss, and chronic fatigue; events that may culminate in life-threatening complications. The pathogenesis of IBD has been characterized as complex/multi-factorial that includes disruption of intestinal epithelial barrier with consequent translocation of commensal microbial products as the prime event that instigates severe immune responses and intestinal inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both male and female will be
* Mild and moderate UC patients diagnosed and confirmed by endoscope

Exclusion Criteria:

* Breast feeding
* Significant liver and kidney function abnormalities
* Colorectal cancer patients
* Patients with severe UC
* Patients taking rectal or systemic steroids
* Patients taking immunosuppressives or biological therapies
* Addiction to alcohol and / or drugs
* Known allergy to the dapagliflozin

Ages: 18 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2028-07-20 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the change in mayo score | 6 months
  The Mayo score is one of the most commonly used disease activity indices in placebo-controlled trials in UC. In its complete form, it is composed of four parts: rectal bleeding, stool frequency, physician assessment, and endoscopy appearance

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt